CLINICAL TRIAL: NCT03400644
Title: Are Rigid Cervical Collars Necessary for Patients Undergoing Open-door Laminoplasty and Titanium Arch Plates for Cervical Myelopathy? - A Randomized Clinical Trial
Brief Title: Are Rigid Cervical Collars Necessary for Open-door Laminoplasty and Titanium Arch Plates for Cervical Myelopathy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Jason Pui Yin Cheung, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: neck_collar1.0
Record Dates: First submitted 2017-12-23; First posted 2018-01-17 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Cervical Myelopathy
Keywords: open-door laminoplasty, laminoplasty, cervical collars

STUDY DESIGN:
Intervention Model Description: Prospective, parallel single-blinded randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Collar (Active Comparator): Subjects are prescribed with custom-made rigid cervical collar which are to be worn for 3 weeks postoperatively
  Interventions: Device: Cervical collar
- Without Collar (No Intervention): Subjects do not need to wear any cervical collar postoperatively

INTERVENTIONS:
Device: Cervical collar — Cervical neck collar which is routinely made for post-laminoplasty patients
  Arms: With Collar

SUMMARY:
This is a randomized controlled trial to assess the use of rigid neck collar postoperatively. It consists of patients with cervical myelopathy undergoing open-door laminoplasty with titanium arch plates. Patients are divided into two groups: one group are not using rigid neck collar whereas the second group of patients wear rigid neck collar for three weeks postoperatively. Both groups of patients will then be assessed at fixed intervals. Clinical assessments include the cervical spine range of motion, any axial neck pain and also a full neurological examination. Radiographs will be used to assess for any complications. Cervical spine alignment and relevant questionnaires will be done and recorded. These results will help to conclude whether we can avoid the use of rigid cervical collars postoperatively, in view of the associated problems arising from restricted neck movement.

DETAILED DESCRIPTION:
Current management protocols regarding cervical laminoplasty is to provide early immobilization with rigid cervical neck collars to avoid implant failure, loss of correction and recurrence of neurological deficit. However, there is no strong evidence supporting the need for neck collars in laminoplasty especially since modern plating fixation methods are already very rigid. Cervical neck collars should also not be used haphazardly due to possible complications and cost implications. Cervical range of motion has been shown to reduce with rigid cervical collars. Decreased voluntary eye movement and postural stability has also been illustrated. Longer duration of neck collar use may even lead to postoperative axial neck pain. Neck collars has also been linked to complications such as pressure ulcers, nerve palsy, skin reactions, dysphagia and respiratory problems. The costs of collar manufacturing and maintenance is not small and must also be taken into consideration. With stronger fixation devices like plates, the above complications can be avoided. Most clinicians still use neck collars for protection mainly due to historical reasons. However this is not an evidence-based approach. By eliminating the need for neck collars, patients are allowed earlier mobilization, less neck stiffness and axial neck pain while reducing its cost. Hence this study is important to provide a basis for changing clinical practice. The study is a prospective randomized controlled trial. Patients are consecutively and randomly divided into two groups . One group of patients will receive no cervical collar postoperatively and a second group will receive rigid neck collar for 3 weeks postoperatively. Operative techniques will be standardized. All assessments are performed 3 and 6 weeks, and 3, 6, 12 and 24 months postoperatively. The subjects were analysed in terms of clinical and functional outcomes through radiographic measurements, clinical assessment and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending either Queen Mary Hospital or Duchess of Kent Children's Hospital, who are over 18 years of age, and present with clinical and radiological signs compatible with cervical myelopathy undergoing laminoplasty. Patients must be literate and able to comprehend the study to be enrolled.

Exclusion Criteria:

* All patients with previous cervical spine surgery, congenital deformities, spine infection or inflammation, tumour, fusion surgery, non-Chinese, undergoing workman's compensation and unable or refuse to follow the standardized rehabilitation protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Cervical spine range of motion (absolute values and changes from baseline, with standard deviations) | 24 months
  To be measured by a single operator using a goniometer
Axial neck pain (absolute values and changes from baseline, with standard deviations) | 24 months
  Patient is asked to rate their axial neck pain on the day of follow-up, with the VAS scale 0-10 with 0 being the least and 10 being the worst pain experienced
SF-36 (absolute values and changes from baseline, with standard deviations) | 24 months
  As a utility score and for assessing any difference between the cervical collar versus the without cervical collar group. The physical health component and mental health component are derived from the following subscales: Physical functioning, role limitations due to physical health, role limitations due to emotional problems, vitality, mental health, social functioning, bodily pain and general health perception
JOA scores (absolute values and changes from baseline, with standard deviations) | 24 months
  JOA consists of 6 domain scores and allow assessment as a composite scores or from individual domain: motor dysfunction in the upper and lower extremities; sensory function in the upper and lower extremities and in the trunk; and the bladder function
Neck Disability Index (absolute values and changes from baseline, with standard deviations) | 24 months
  An outcome score in assessing how neck pain affecting subjects' daily life activities
Spinal canal diameters at C3, C4, C5, C6 | 24 months
  To measure any difference between 2 study groups at various time points

SECONDARY OUTCOMES:
Rate of recovery (in percentage) | 24 months
  to be derived from the JOA scores

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong